CLINICAL TRIAL: NCT06219434
Title: Pilot Feasibility Evaluation of a Mindfulness (Mindfulness) Intervention in Women Preparing for Chemotherapy for Breast Cancer
Brief Title: Evaluation of a Mindfulness Intervention to Prevent Chemo-brain in Women Preparing for Chemotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: iRISID-2023-2430; JT 32145 (Other: JeffTrial Number)
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness; Mindfulness-Based Stress Reduction; Specimen Handling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (mindfulness program) (Experimental): Patients participate in a mindfulness program composed of topics that include mindfulness of breathing and the body scan, mindful eating, mindful activity, mindfulness in daily life, expanding the field of awareness, and maintaining a flexible mindfulness practice weekly over 2.5 hours for 8 weeks. Patients also undergo blood sample collection and fMRI on the study.
  Interventions: Behavioral: Mindfulness Relaxation; Procedure: Functional Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Mindfulness Relaxation — Participate in mindfulness program
  Other Names: MBSR; Mindful Meditation; Mindfulness Meditation; Mindfulness-Based Stress Reduction
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI
  Other Names: fMRI; FUNCTIONAL MRI
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well a mindfulness intervention helps the prevention of chemotherapy-brain (chemo-brain) in women preparing for chemotherapy for breast cancer. Cognitive dysfunction after chemotherapy has been well-documented. Factors that have been used to document and/or have been correlated with chemo brain include self-report and structural brain changes including volume loss. Mindfulness is a type of meditation practice that can be learned to support well-being and decrease stress. Mindfulness is an approach that helps the person increase their awareness of the present moment without judgement. There are data that mindfulness may increase attention and concentration which may prevent some of the side effects from chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of an 8-week mindfulness intervention in women preparing for chemotherapy for breast cancer.

II. Evaluate cognitive dysfunction related factors as an exploratory objective: cognitive function, quality of life, inflammatory markers, functional magnetic resonance imaging (fMRI) brain imaging, and a record of mindfulness practice.

OUTLINE:

Patients participate in a mindfulness program composed of topics that include mindfulness of breathing and the body scan, mindful eating, mindful activity, mindfulness in daily life, expanding the field of awareness, and maintaining a flexible mindfulness practice weekly over 2.5 hours for 8 weeks. Patients also undergo blood sample collection and fMRI on the study.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Breast cancer diagnosis preparing to undergo chemotherapy

Exclusion Criteria:

* Under the age of 18
* Cannot provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Participation rate | Up to 1 year
  Will be determined by 75% of the participants will participate in at least 6 of the 8 mindfulness sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hopsital, Philadelphia, Pennsylvania, United States